CLINICAL TRIAL: NCT05368935
Title: An Open-label, Phase 1, Multiple-dose Study to Evaluate the Pharmacokinetics of Nitazoxanide 500 mg Twice Daily for 7 Days in Adult Subjects With Mild, Moderate, and Severe Renal Impairment and Adult Healthy Control Subjects
Brief Title: Nitazoxanide Pharmacokinetic Parameters in Renal Impaired Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NTZ-122-1
Record Dates: First submitted 2022-04-12; First posted 2022-05-10 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Renal Impairment; Renal Disease; Kidney Disease
Keywords: Pharmacokinetics; Healthy Volunteer; Renal Disease; Kidney Disease; Renal Impairment; Antiparasitic; Antiprotozoal
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases | interventions — nitazoxanide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Control Match (RF ≥ 90 mL/min) (Experimental): 500 mg Twice Daily for 7 days
  Interventions: Drug: Nitazoxanide
- Mild Renal Impairment (RF ≥ 60 to < 90 mL/min) (Experimental): 500 mg Twice Daily for 7 days
  Interventions: Drug: Nitazoxanide
- Moderate Renal Impairment (RF ≥ 30 to < 60 mL/min) (Experimental): 500 mg Twice Daily for 7 days
  Interventions: Drug: Nitazoxanide
- Severe Renal Impairment (RF < 30 mL/min and not on dialysis) (Experimental): 500 mg Twice Daily for 7 days
  Interventions: Drug: Nitazoxanide

INTERVENTIONS:
Drug: Nitazoxanide — 500 mg Twice Daily for 7 days
  Other Names: NTZ

SUMMARY:
This study is being conducted to evaluate the major Nitazoxanide (NTZ) active metabolite in adult participants with renal impairment and healthy adults.

DETAILED DESCRIPTION:
This study is being conducted to assess the pharmacokinetics of the major Nitazoxanide active metabolite as well as the safety and tolerability in renal impaired (mild, moderate and severe) and healthy matched control adults following repeated oral dose administration of NTZ 500 mg twice a day for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, between 18 and 80 years of age, inclusive
2. With a minimum body weight of ≥ 50.0 kg for males and ≥ 45.0 kg for females and within a BMI range of 18.0 to 40.0 kg/m^2, inclusive
3. Females participating in this study must be of non-childbearing potential or must be using highly effective contraception for the full duration of the study
4. Matched to subjects with mild, moderate and/or severe renal impairment in age (± 15 years), BMI (± 20%) and sex
5. The diagnosis of renal impairment has been stable, without significant change in overall disease status in the last 3 months prior to screening

Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

1. Positive serum pregnancy test at screening or positive urine pregnancy test
2. Having taken NTZ at any time prior to the first study drug administration
3. History of alcohol abuse within 1 year prior to screening
4. History of drug abuse within 1 year prior to screening or recreational use of soft drugs within 1 month or hard drugs within 3 months prior to screening
5. Excessive consumption of xanthine-based drinks (> 4 cups or glasses per day), food or beverages containing xanthine derivatives or xanthine-based compounds, 48 hours prior to the first dosing
6. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to the first dosing
7. Strenuous exercise within 72 hours prior to check-in
8. History of a major surgical procedure within 30 days prior to screening
9. Presence or history of malignancy within the prior 3 years, with the exception of treated basal cell or squamous cell carcinoma
10. Poor peripheral venous access
11. Subjects who are taking warfarin or other highly plasma protein-bound drugs with narrow therapeutic indices

Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18; 24 hours (Day 8); 48 hours (Day 9); 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetic (PK) parameters of NTZ active metabolite expressed in terms of unbound as well as total concentrations at steady-state in subjects with mild, moderate and severe renal impairment compared to healthy volunteers
Area under the plasma concentration time curve (AUC) from time zero to the time of the last quantifiable concentration (AUC0-t) | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18; 24 (Day 8); 48 (Day 9); 72 (Day 10) and 96 (Day 11) hours post-dose
  Plasma pharmacokinetic parameters of NTZ active metabolite expressed in terms of unbound as well as total concentrations at steady-state in subjects with mild, moderate and severe renal impairment compared to healthy volunteers
AUC from time zero to 12h (AUC0-12) | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18; 24 hours (Day 8); 48 hours (Day 9); 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetic parameters of NTZ active metabolite expressed in terms of unbound as well as total concentrations at steady-state in subjects with mild, moderate and severe renal impairment compared to healthy volunteers

SECONDARY OUTCOMES:
Time of the maximum observed plasma concentration (Tmax) for NTZ and its major active metabolite | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18 hours; 24 hours (Day 8); 48 hours (Day 9) ; 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetics
Apparent plasma terminal elimination half-life (t1/2) for the NTZ and its major active metabolite | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18 hours; 24 hours (Day 8); 48 hours (Day 9) ; 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetics
Unbound fraction in plasma defined as total concentration/unbound concentration (fu) for the NTZ and its major active metabolite | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18 hours; 24 hours (Day 8); 48 hours (Day 9) ; 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetics
Area under the plasma concentration-time curve from time zero to infinity (extrapolated) (AUC0-∞) for the NTZ and its major active metabolite | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18 hours; 24 hours (Day 8); 48 hours (Day 9) ; 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetics
Trough concentration (Ctrough) for the NTZ and its major active metabolite | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18 hours; 24 hours (Day 8); 48 hours (Day 9) ; 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetics
Cmax for the NTZ major active metabolite | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18 hours; 24 hours (Day 8); 48 hours (Day 9) ; 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetics
AUC0-12 for the NTZ major active metabolite | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18 hours; 24 hours (Day 8); 48 hours (Day 9) ; 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetics
AUC0-t for the NTZ major active metabolite | Day 1: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10 and 12 hours post dose; Day 2-6: pre-dose; Day 7: pre-dose; 1; 2; 3; 4; 5; 6; 7; 8; 10; 12; 14; 16; 18 hours; 24 hours (Day 8); 48 hours (Day 9) ; 72 hours (Day 10) and 96 hours (Day 11) post-dose
  Plasma pharmacokinetics
Amount of drug excreted in urine over the time interval between t1 and t2 (Aet1-t2) for the NTZ major active metabolites | Day (D) 1: pre-dose, 0-4 hours (h); 4-8 h; and 8-12 h post-morning dose; D7: 0-4 h; 4-8 h; 8-12 h; 12- 24 h; 24-48 h; 48-72 h and 72-96 h post-dose
  Urine pharmacokinetics
Cumulative amount of drug excreted in urine from time zero until and up to infinity (Ae0-∞) for the NTZ major active metabolites | Day (D) 1: pre-dose, 0-4 hours (h); 4-8 h; and 8-12 h post-morning dose; D7: 0-4 h; 4-8 h; 8-12 h; 12- 24 h; 24-48 h; 48-72 h and 72-96 h post-dose
  Urine pharmacokinetics
Cumulative amount of drug excreted in urine from time zero until the last measured concentration at time t (Ae0-t) for the NTZ major active metabolites | Day (D) 1: pre-dose, 0-4 hours (h); 4-8 h; and 8-12 h post-morning dose; D7: 0-4 h; 4-8 h; 8-12 h; 12- 24 h; 24-48 h; 48-72 h and 72-96 h post-dose
  Urine pharmacokinetics
Percentage of dose excreted in urine over the time interval between t1 and t2 (Fet1-t2) for the NTZ major active metabolites | Day (D) 1: pre-dose, 0-4 hours (h); 4-8 h; and 8-12 h post-morning dose; D7: 0-4 h; 4-8 h; 8-12 h; 12- 24 h; 24-48 h; 48-72 h and 72-96 h post-dose
  Urine pharmacokinetics
Cumulative percent of dose excreted in urine from time zero until the last measured concentration at time t (Fe0-t) for the NTZ major active metabolites | Day (D) 1: pre-dose, 0-4 hours (h); 4-8 h; and 8-12 h post-morning dose; D7: 0-4 h; 4-8 h; 8-12 h; 12- 24 h; 24-48 h; 48-72 h and 72-96 h post-dose
  Urine pharmacokinetics
Renal clearance (CLR) for the NTZ major active metabolites | Day (D) 1: pre-dose, 0-4 hours (h); 4-8 h; and 8-12 h post-morning dose; D7: 0-4 h; 4-8 h; 8-12 h; 12- 24 h; 24-48 h; 48-72 h and 72-96 h post-dose
  Urine pharmacokinetics
Cmax after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
AUC0-12 after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
AUC0-t after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
AUC0-∞ after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
Tmax after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
t1/2 after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
Aet1-t2 after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
Amount of drug excreted in urine from time zero to 12h (Ae0-12) after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
Fet1-t2 after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
Cumulative percent of dose excreted in urine from time zero to 12h (Fe0-12) after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics
CLR after the single oral administration of NTZ 500 mg for the NTZ major active metabolites | D1:predose;1;2;3;4;5;6;7;8;10;12h post dose; D2-6:predose; D7:predose;1;2;3;4;5;6;7;8;10;12;14;16;18; 24(D8);48(D9);72(D10) and 96(11)h post-dose.Urine:D1 predose; 0-4; 4-8; 8-12 h post morning dose; D7 0-4;4-8;8-12;12- 24;24-48;48-72;72-96h post-dose
  Plasma and urine pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Carol Addy, MD, Study Director — Genfit
Locations (2):
- United States (2):
  - Panax Clinical Research, Miami Lakes, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No